CLINICAL TRIAL: NCT04000750
Title: The Influence of 16:8 Time-Restricted Eating on Resistance Exercise-Induced Skeletal Muscle Hypertrophy
Brief Title: Time-Restricted Eating and Muscle Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Fullerton (Other)
Collaborators: San Francisco State University (Other)
Responsible Party: Principal Investigator, Andrew Galpin, Associate Professor, California State University, Fullerton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSP Fullerton
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Muscle Hypertrophy; Healthy and Well-Trained Men and Women
Keywords: Hypertrophy; Intermittent Fasting; Time Restricted Eating; Protein Signaling; Anabolic
MeSH Terms: conditions — Hypertrophy; Intermittent Fasting | interventions — Resistance Training; Whey Proteins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will know their group. Training and Nutrition research team members will know the participants group. Data analysis team will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (16:8) (Experimental): Participants will consume all calories within an 8 hour window each day.
  Interventions: Other: Time Restricted Eating; Other: Resistance Training; Dietary Supplement: Whey Protein
- Control (Active Comparator): Participants will consume all calories within a ~12 hour window each day (4 separate meals + needed snacks).
  Interventions: Other: Normal Feeding; Other: Resistance Training; Dietary Supplement: Whey Protein

INTERVENTIONS:
Other: Time Restricted Eating — Diet will be tracked and reported every day to a qualified dietitian.
  Arms: Time Restricted Eating (16:8)
Other: Normal Feeding — Diet will be tracked and reported every day to a qualified dietitian.
  Arms: Control
Other: Resistance Training — 8 weeks of supervised and programmed whole body resistance training, performed 4x per week
Dietary Supplement: Whey Protein — Consumed on all exercise days.

SUMMARY:
The purpose is to examine the effects of time-restricted eating (TRE; consuming all calories within an 8-hour period each day) vs. normal eating (CON; consuming same kcals and protein as TRE, but during a 10-13 hr eating window each day) during 8 weeks of resistance exercise on body composition and muscle mass (whole muscle and single fiber), muscular performance, anabolic protein signaling, single muscle fiber characteristics, and the gut microbiome in well-trained young men and women.

DETAILED DESCRIPTION:
The primary goal pertains to muscle hypertrophy (not fat loss), thus all participants will be placed in a 10% caloric surplus.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old with <25% (men) or <30% (women) body fat
* have experience in resistance exercise for the whole body and performed resistance exercise at least 3 times per week the last 12 months
* be able to perform all necessary exercises with safe technique and no pain
* be able to squat 1.5x (men) or 1x (women) body weight
* be able to bench press 1.1x (men) or 0.55x (women) body weight
* be on a non-specialized, mixed macronutrient diet
* have a lifestyle which enables a reasonably consistent 7+ hours of sleep per night
* be free of any current joint, musculoskeletal, and/or neuromuscular injuries

Exclusion Criteria:

* have any known current illness, prohibitive muscular or neuromuscular problem, hypertension, cardiac, pulmonary, liver, kidney, insulin or any other metabolic disorders (e.g. Type I or Type II diabetes)
* are lactose intolerant or unable to consume whey protein for any reason
* are on any medications known to affect protein metabolism
* have taken antibiotics in the last 6 months
* cannot refrain from consuming any alcoholic beverages, nicotine, or marijuana (or derivative) for a period of 48 hours prior to data collection (pre and post testing)
* consume alcohol >2x per week
* consume any analgesic or anti-inflammatory drug(s), prescription or non-prescription, chronically or within 48 hours of data collection
* consume any recreational drug(s), prescription or non-prescription, legal or illegal, chronically or within 30 days of data collection
* consume any caffeine or food within 12 hours of data collection
* cannot refrain from physical exercise (outside of activities of daily living) outside of what is prescribed by the research team for the duration of the study
* cannot refrain from using recovery methods such as electric stimulation, hot/cold therapy, massage, chiropractic, or personal air/water devices (Normatech, etc.)
* have utilized any anabolic steroid, currently or in the past
* cannot refrain from consumption of any supplementation (creatine, multivitamin, fish oil, protein powder, BCAA, pre-workouts, etc.) outside of what is provided
* cannot refrain from consuming any supplemental pro or prebiotics or other items that intentionally alter the gut microbiome
* fail to adhere to the nutritional guidelines or miss >3 of the exercise sessions
* were recently pregnant, trying to become pregnant, or are currently breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Changes in Muscle Size - Lower Body | Pre, Mid (4 weeks), and Post (8 weeks)
  via Ultrasound
Changes in Muscle Size - Upper Body | Pre, Mid (4 weeks), and Post (8 weeks)
  via Ultrasound
Changes in Fiber Type-Specific Size | Pre and Post (week 8)
  Single muscle fiber analysis
Changes in Body composition | Pre, Mid (4 weeks), and Post (8 weeks)
  via BodPod
Acute Exercise Induced Fiber Type-Specific Anabolic Signaling (Total Concentration and Phosphorylation Status) | Day 1 of exercise training
  Men only; assessed via single fiber Simple Western

SECONDARY OUTCOMES:
Changes in Maximal Strength | Pre and Post (week 8)
  1RM on bench press, squat, and leg extension
Changes in Maximal Muscular Endurance | Pre and Post (week 8)
  Maximal repetitions on bench press and leg press
Changes in Gut Microbiome | Pre, Mid (week 2, 4, 6), and Post (week 8)
  via stool sample
Changes in Fiber Type Composition | Pre and Post (week 8)
  Single Fiber via SDS-PAGE
Changes in Fiber Type-Specific Resting Anabolic Signaling (Total Concentration and Phosphorylation Status) | Pre and Post (week 8)
  via single fiber Simple Western
Changes in Mood | Weekly for duration of the intervention (8 weeks)
  via Questionnaire
Changes in Enjoyment of Diet | Weekly for duration of the intervention (8 weeks)
  via Questionnaire
Changes in Sleep (total and quality) | Weekly for duration of the intervention (8 weeks)
  via Questionnaire
Changes in Menstrual Cycle | Pre, Mid (week 4), and post (week 8)
  via Questionnaire; women only
Total Training Volume | After 8 weeks
Nutrient Intake | Daily, starting 7 days before the study and continuing for 8 additional weeks
  Total Kcal and grams of protein, fat, and carbohydrates

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sport Performance at California State University, Fullerton, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No